CLINICAL TRIAL: NCT00279110
Title: Directly Administered vs. Self-administered Antiretroviral Therapy in Methadone Clinics
Brief Title: Directly Administered HIV Therapy in Methadone Clinics
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Gregory M. Lucas, MD PhD, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA018577 (NIH)
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2011-05

CONDITIONS: HIV Infections; Heroin Dependence
Keywords: HIV; Antiretroviral therapy; Heroin dependence; Methadone; Buprenorphine
MeSH Terms: conditions — HIV Infections; Heroin Dependence

ARMS (2):
- A (Experimental)
  Interventions: Behavioral: Directly administered antiretroviral therapy (DAART)
- B (No Intervention)

INTERVENTIONS:
Behavioral: Directly administered antiretroviral therapy (DAART) — Participants are observed taking HIV medications on days when they receive opioid agonist therapy.
  Arms: A

SUMMARY:
The purpose of this study is to determine whether providing directly administered antiretroviral therapy to HIV-infected who receive methadone therapy leads to better treatment outcomes than if they take HIV medications on their own.

DETAILED DESCRIPTION:
We propose to conduct a randomized, unblinded, clinical trial of a medication adherence intervention in opioid-dependent, HIV-infected participants who are initiating new antiretroviral therapy, and who receive opioid agonist maintenance therapy with methadone or buprenorphine in opioid treatment programs (OTPs) in Baltimore, MD. Randomization will be stratified by study site and prior antiretroviral exposure. Two hundred participants will be randomly assigned 1:1 self-administered antiretroviral therapy (SAT) or directly administered antiretroviral therapy (DAART). Subjects assigned to DAART will take morning doses of antiretroviral therapy with a nurse or medical assistant in a private room at the OTP. DAART subjects will be transferred to self-administered therapy after 12 months. This is a 5 year study and participants will be enrolled between month 6 and month 42 of the study. The maximum follow-up for individual participants will be 18 months. Based on our pilot experience we anticipate 50% of subjects will be women, 80% African American, with a median age of 44 years. The following outcomes will be compared in the two study arms:

* Suppression of the viral load (primary outcome)
* Changes in CD4+ cell counts
* The development of antiretroviral drug resistance
* Retention to opioid agonist maintenance therapy, urine toxicology screens for drugs of abuse, and self-reported drug and alcohol use
* Self-reported adherence with therapy, retention to ART, and clinical and psychosocial moderators of adherence
* Electronically monitored medication adherence, using MEMS caps, in the first 2 months of the study

Outcomes data will be obtained at study assessment visits at baseline, 3 months, 6 months, 12 months, and 18 months. Participants will provide contact information, take an interviewer-administered survey, and provide blood and urine samples at study assessment visits. MEMS cap data will be captured at 1 month and 2 months. Subjects will be compensated for successful completion of study assessment visits and MEMS interrogations.

ELIGIBILITY:
Inclusion Criteria:

1. Eighteen years of age or older
2. Documented serologic evidence of HIV infection (positive ELISA and Western blot)
3. Identifiable medical provider, who is responsible for managing HIV treatment
4. Proof that ART has been prescribed and that patient has prescription medication coverage
5. Nadir CD4+ cell count < 350/mm3 or off-treatment HIV RNA > 55,000 copies/ml if asymptomatic and ART naive
6. Current plasma HIV RNA > 500 copies/ml
7. Initiating ART for first time, reinitiating therapy after stopping, or changing therapy due to virologic failure
8. ART with at least 3 agents, including a protease inhibitor, a non-nucleoside reverse transcriptase inhibitor, or abacavir
9. Methadone or buprenorphine maintenance therapy > 3 weeks, with no planned detoxification

Exclusion Criteria:

1. Need to use ART dosed more frequently than twice daily,
2. Need to use a liquid preparation of antiretroviral medication,
3. Documented triple-class antiretroviral resistance (defined below),
4. Participation in another study or program that includes directly observed therapy.
5. Use of ART regimens that are expressly discouraged in DHHS HIV clinical care guidelines

Triple-class antiretroviral resistance will be defined according to IAS-USA interpretive guidelines: NRTI class - 3 thymidine or non-thymidine-associated mutations (excluding the M184V mutation) or a multi-nucleoside resistance mutation in reverse transcriptase; PI class - 3 protease mutations, including 1 primary mutation; NNRTI class - 1 primary (K103N or Y188L) or 2 secondary NNRTI-associated mutations in reverse transcriptase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2006-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
HIV RNA < 50 c/mL | 12 months

SECONDARY OUTCOMES:
Log10 change in HIV RNA from baseline | 12 months
HIV RNA < 50 c/mL 6 mos. after intervention | 18 months
Log10 change in HIV RNA from baseline 6 months post intervention | 18 months
Change in CD4 cell count from baseline | 18 months
ART utilization | 12 months
Development of antiretroviral resistance | 12 months
Retention to substance abuse treatment | 12 months
Urine drug screen positivity in follow-up | 12 months
Electronically monitored adherence | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Gregory M. Lucas, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (5):
- United States (5):
  - Baltimore VA Drug Dependency Program, Baltimore, Maryland
  - Program for Alcohol and Other Drug Dependencies, Baltimore, Maryland
  - Man Alive, Inc., Baltimore, Maryland
  - New Hope Treatment Center, Baltimore, Maryland
  - Day Break Methadone Clinic, Baltimore, Maryland

REFERENCES:
- [Background] Mullen BA, Cook K, Moore RD, Rand C, Galai N, McCaul ME, Glass S, Oursler KK, Lucas GM. Study design and participant characteristics of a randomized controlled trial of directly administered antiretroviral therapy in opioid treatment programs. BMC Infect Dis. 2011 Feb 15;11:45. doi: 10.1186/1471-2334-11-45. PMID 21324133
- [Result] Lucas GM, Mullen BA, Galai N, Moore RD, Cook K, McCaul ME, Glass S, Oursler KK, Rand C. Directly administered antiretroviral therapy for HIV-infected individuals in opioid treatment programs: results from a randomized clinical trial. PLoS One. 2013 Jul 16;8(7):e68286. doi: 10.1371/journal.pone.0068286. Print 2013. PMID 23874575